CLINICAL TRIAL: NCT00254917
Title: Assessment of the Immunogenicity and Safety of PENTAXIM™ in Philippines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E2I29
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Diphtheria; Tetanus; Polio; Pertussis; Haemophilus Influenzae Type B
Keywords: Pentaxim
MeSH Terms: conditions — Diphtheria; Tetanus; Poliomyelitis; Whooping Cough; Haemophilus Infections | interventions — Tetanus Toxoid; HibTITER protein, Haemophilus influenzae; Pentavac

ARMS (2):
- 1 (Experimental): Concommitant recombinant hepatitis B vaccine at 0, 6 and 14 weeks of age
  Interventions: Biological: Diphteria, Tetanus, Polio, Acellular Pertussis, Hib vaccine
- 2 (Experimental): Concommitant recombinant hepatitis B vaccine at 6, 10, and 14 weeks of age.
  Interventions: Biological: Diphteria, Tetanus, Polio, Acellular Pertussis, Hib vaccine

INTERVENTIONS:
Biological: Diphteria, Tetanus, Polio, Acellular Pertussis, Hib vaccine — 0.5 mL, IM
  Other Names: PENTAXIM™
  Arms: 1
Biological: Diphteria, Tetanus, Polio, Acellular Pertussis, Hib vaccine — 0.5 mL, IM
  Other Names: PENTAXIM™
  Arms: 2

SUMMARY:
The present clinical study will assess the immunogenicity and reactogenicity of the subsequent administration of Aventis Pasteur's DTacP-IPV//PRP~T combined vaccine (PENTAVAC™/PENTAXIM), as a three-dose primary vaccination in 6, 10 and 14 weeks of age schedule followed by a booster vaccination during the second year of life with the aim to cover the WHO EPI primary vaccination schedule at this age for diphtheria, tetanus, pertussis, poliomyelitis and Hib vaccines.

WHO EPI vaccination schedules for hepatitis B (either 0, 6 and 14 weeks or 6, 10 and 14 weeks of age) will be also assessed in infants born to HBsAg seronegative mothers.

To assess the safety of Pentaxim.

DETAILED DESCRIPTION:
Open, randomized, multicentric, controlled trial. Infants will be randomly allocated in one of the two study groups as follows:

Group A: 212 subjects will receive the PENTAXIM™ vaccine at 6, 10 and 14 weeks of age, and the recombinant 10 µg hepatitis B vaccine at 0, 6 and 14 weeks of age.

Group B: 212 subjects will receive the PENTAXIM™ and the recombinant 10 µg hepatitis B vaccines at 6, 10 and 14 weeks of age.

All infants included in the study will receive a booster dose of PENTAXIM™ vaccine at 18-19 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by one or both parent(s) and/or by a legally accepted representative prior to the first study intervention
* Healthy male or female newborn
* Age ranging from birth to 48 hours of life (included)
* Birth weight >2.5 kg and gestational age >37 weeks
* Born to HBs antigen-negative mother

Exclusion Criteria:

* Known previous therapy of the mother with cadaveric pituitary derived human growth hormone
* Infant presently enrolled or scheduled to be enrolled in another clinical trial
* Infant with moderate or severe illness, mainly infectious diseases
* Infant with fever (rectal temperature > 38°C or axillary temperature > 37.5°C)
* Infant with severe congenital defects or abnormalities
* Uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection.
* Known immunological deficiency (including a known HIV seropositive mother)
* Administration of vaccine since birth (other than BCG)
* Previous or planned administration of immunosuppressive therapy, immunoglobulins and /or any blood-derived products (inhaled and topical corticoids are allowed)

Ages: 6 Weeks to 19 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 387 (Actual)
Dates: Start 2003-10; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the safety of PENTAXIM™ Vaccine. | 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Manila, Philippines

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com